CLINICAL TRIAL: NCT01783249
Title: The Influence of Exercise on Anemia in MDS Patients
Brief Title: Influence of Exercise on Anemia in MDS Patients
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: We were unable to find patients that fit the eligibility criteria.
Sponsor: University of Rochester (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 37173MDS
Record Dates: First submitted 2011-11-30; First posted 2013-02-04 (Estimated); Last update posted 2013-02-04 (Estimated); Status verified 2013-01

CONDITIONS: Feasibility Pilot Study

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): Usual care monitoring
- Exercise using stationary cycling (Other): Stationary cycling exercise program
  Interventions: Other: Stationary Exercise cycling

INTERVENTIONS:
Other: Stationary Exercise cycling — Stationary exercise cycling
  Arms: Exercise using stationary cycling

SUMMARY:
That exercise will reduce anemia and fatigue, while improving aerobic capacity, strength and hematopoietic stem and progenitor cell mitochondrial function.

ELIGIBILITY:
Inclusion Criteria:Have a confirmed diagnosis of MDS, Have approval of the study medical monitor, be able to read English, be 21 years of age or older, give informed consent -

Exclusion Criteria: Have physical limitations, be identified in the active or maintenance stage of exercise behavior

-

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-11; Primary Completion 2012-11 (Estimated); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Feasibility data on the effect of a stationary cycling program
  Aim to provide preliminary feasibility data on the effect of a stationary cycling program on anemia and acrocytosis, fatigue, aerobic capacity, strength, and hematopoietic stem and progenitor cell mitochondrial function in MDS patients.

CONTACTS AND LOCATIONS:
Locations (1):
- James P. Wilmot Cancer Center, University of Rochester, Rochester, New York, United States